CLINICAL TRIAL: NCT00594230
Title: A Phase II Trial of LBH589 in Refractory Myelodysplastic Syndromes (MDS) Patients
Brief Title: LBH589 in Refractory Myelodysplastic Syndromes (MDS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Per protocol, the results of a planned interim analysis demonstrated insufficient efficacy and led to early termination of the study.
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRI MDS 07
Record Dates: First submitted 2007-12-19; First posted 2008-01-15 (Estimated); Results first posted 2012-12-19 (Estimated); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Myelodysplastic Syndromes (MDS)
Keywords: Myelodysplastic Syndromes (MDS); Refractory; LBH589
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Panobinostat 20 mg (Experimental): Treatment with LBH589 (Panobinostat) 20 mg
  Interventions: Drug: Panobinostat
- Panobinostat 30 mg (Experimental): Treatment with LBH589 (Panobinostat) 30 mg
  Interventions: Drug: Panobinostat

INTERVENTIONS:
Drug: Panobinostat — Panobinostat(20 mg or 30 mg PO) will be administered three times a week on Monday, Wednesday and Friday. Treatment will be given over 21 days followed by a 7 day rest period and repeated every 28 days. Patients will be assessed for toxicity on an ongoing basis and disease assessment will be determined every 2 treatment cycles (8 weeks). Patients will be allowed to continue on treatment for a maximum of eight four week treatment cycles. Treatment will be discontinued if there is evidence of disease progression, unacceptable toxicity and/or at the discretion of the investigator.
  Other Names: LBH589

SUMMARY:
This will be a single arm Phase II study.

DETAILED DESCRIPTION:
LBH589 (20 mg PO) will be administered three times a week on Monday, Wednesday and Friday. Treatment will be given over 21 days followed by a 7 day rest period and repeated every 28 days. Patients will be assessed for toxicity on an ongoing basis and disease assessment will be determined every 2 treatment cycles (8 weeks). Patients will be allowed to continue on treatment for a maximum of eight four week treatment cycles. Treatment will be discontinued if there is evidence of disease progression, unacceptable toxicity and/or at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytological documented diagnosis of myelodysplastic syndrome (MDS).
* Male or female patients aged >= 18 years old.
* MDS patients who have failed hypomethylating (azacitidine or decitabine) therapy.
* Patients with 5q-cytogenic abnormalities must also have progressed on or been intolerant to lenalidomide.
* Patients with up to and including 30% blasts (FAB RAEB-T) will be eligible to enroll.
* CMML with >= 5% blasts will be eligible to enroll.
* ECOG PS 0, 1 or 2.
* Laboratory values must be as follows:

Bilirubin <= 1.5 mg/dL AST/SGOT <= 2.5 x ULN ALT/SGPT Creatinine <= 2.0 mg/dL or 24-hour Creatinine Clearance >= 50 ml/min Albumin >= 3 g/dL Potassium >= lower limit normal (LLN) Phosphorous >= LLN Calcium >= LLN Magnesium >= LLN

* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to start of treatment.
* Life expectancy >= 12 weeks.

Exclusion Criteria:

* Prior treatment with an HDAC inhibitor.
* Prior intensive chemotherapy or high dose ara-C (>= 1 gm/m2)
* More than one prior single agent chemotherapy regimen. Prior hydroxyurea for cytoreduction will be permitted however.
* Impaired cardiac function
* Active CNS disease, including leptomeningeal metastases.
* Unresolved diarrhea > CTCAE grade 1.
* Chemotherapy, investigational drug therapy, major surgery < 4 weeks prior to starting study drug or patients that have not recovered from side effects of previous therapy.
* Patient is < 5 years free of another primary malignancy except if the other primary malignancy is not currently clinically significant or requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed.
* Women who are pregnant or breast feeding or women of childbearing potential (WOCBP) not willing to use a double barrier method of contraception during the study and 3 months after the end of treatment. One of these methods of contraception must be a barrier method.
* Male patients whose sexual partners are WOCBP not using a double method of contraception during the study and 3 months after the end of treatment. One of these methods must be a condom.
* Patients with gastrointestinal (GI) tract disease, causing the inability to take oral medication, malabsorption syndrome, a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis).
* Other concurrent severe, uncontrolled systemic fungal, bacterial, viral or other infection or intercurrent illness, including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with uncontrolled coagulopathy.
* Abnormal thyroid function (TSH or free T4) detected at screening. Patients with known hypothyroidism who are stable on thyroid replacement are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian W. Flinn, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (7):
- United States (7):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Oncology Hematology Care, Cincinnati, Ohio
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Panobinostat 30 mg: Panobinostat(30 mg PO) will be administered three times a week on Monday, Wednesday and Friday. Treatment will be given over 21 days followed by a 7 day rest period and repeated every 28 days. Patients will be assessed for toxicity on an ongoing basis and disease assessment will be determined every 2 treatment cycles (8 weeks). Patients will be allowed to continue on treatment for a maximum of eight four week treatment cycles. Treatment will be discontinued if there is evidence of disease progression, unacceptable toxicity and/or at the discretion of the investigator.
- Panobinostat 20 mg: Panobinostat(20 mg PO) will be administered three times a week on Monday, Wednesday and Friday. Treatment will be given over 21 days followed by a 7 day rest period and repeated every 28 days. Patients will be assessed for toxicity on an ongoing basis and disease assessment will be determined every 2 treatment cycles (8 weeks). Patients will be allowed to continue on treatment for a maximum of eight four week treatment cycles. Treatment will be discontinued if there is evidence of disease progression, unacceptable toxicity and/or at the discretion of the investigator.
Period: Overall Study
Arm/Group | Panobinostat 30 mg | Panobinostat 20 mg
Started | 16 | 10
Completed | 1 | 1
Not Completed | 15 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panobinostat 30 mg | Panobinostat 20 mg | Total
Number analyzed (Participants) | 16 | 10 | 26
Age, Continuous [Median (Full Range); unit: years] | 75 [59 to 86] | 74 [64 to 84] | 75 [59 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7
  Male | 15 | 4 | 19
Region of Enrollment [Number; unit: participants]
  United States | 16 | 10 | 26

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (CR, Marrow CR + PR) of LBH in Patients With Relapsed or Refractory MDS.
Description: Overall response rate (ORR) is defined by the modified International Working Group (IWG) Response Criteria for MDS. In the marrow, Complete Response (CR) is <= 5% blasts present with normal maturation of all cell lines. In peripheral blood, CR is defined as hemoglobin >= 11 g/dL, ANC >= 1000/mL, and platelets >= 100,000 with 0% blasts present. Partial Response (PR) is defined the same as CR with blasts decreased by >= 50% and >= 5% blasts in the marrow.
Time Frame: Every 8 weeks up to 24 months on-study.
Population: All evaluable patients assessed for response prior to early study termination - one patient in each arm was not evaluable due to coming off-study prior to assessment
Measure: Number; unit: participants
Arm/Group | Panobinostat 30 mg | Panobinostat 20 mg
Number analyzed (Participants) | 15 | 9
participants | 0 | 0

2. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression is defined as the time between day 1 cycle 1 and time to first documented disease progression. Disease progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Every 8 weeks up to 24 months on-study, every 3 months in follow-up until progression of disease
Population: Study terminated early, no results are available for this endpoint as the analysis was not done.
Arm/Group | Panobinostat 30 mg | Panobinostat 20 mg
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Hematologic Improvement, Including Transfusion Independence
Description: Hematologic measures will include total WBC and platelets
Time Frame: Every 8 weeks up to 24 months on-study
Population: Study terminated early, no results are available for this endpoint as the analysis was not done
Arm/Group | Panobinostat 30 mg | Panobinostat 20 mg
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from when objective response is realized until time to first documented disease progression. Disease progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Objective Response = CR + PR. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Every 8 weeks up to 24 months on-study
Population: Study terminated early, no results are available for this endpoint as the analysis was not done
Arm/Group | Panobinostat 30 mg | Panobinostat 20 mg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Median Time to Treatment Failure
Description: Time to treatment failure is defined as measuring the time between cycle 1 day 1 to discontinuation for any reason.
Time Frame: 24 months
Population: Study terminated early, no results are available for this endpoint as the analysis was not done
Arm/Group | Panobinostat 30 mg | Panobinostat 20 mg
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Median Overall Survival
Description: The Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Death
Time Frame: 24 months on-study, patients followed every 3 months in follow-up
Population: Study terminated early, no results are available for this endpoint as the analysis was not done
Arm/Group | Panobinostat 30 mg | Panobinostat 20 mg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Safety and Tolerability of LBH589 in Patients With Relapsed/Refractory MDS by Measuring the Number of Participants With Adverse Events
Description: The reported incidence of AEs and SAEs with an onset on or after the initiation of therapy was graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat 30 mg | Panobinostat 20 mg
Number analyzed (Participants) | 16 | 10
Participants | 15 | 9

ADVERSE EVENTS:
Arm/Group | Panobinostat 20 mg | Panobinostat 30 mg
Serious Adverse Events (participants affected / at risk) | 3/10 | 6/16
Other Adverse Events (participants affected / at risk) | 9/10 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panobinostat 20 mg (N=10) | Panobinostat 30 mg (N=16)
Abdominal Pain (Gastrointestinal disorders) | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 4
Infections and infestations - Other, pneumonia (Infections and infestations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Pain (General disorders) | 0 | 1
General disorders and administration site conditions - Other, compartment syndrome (General disorders) | 0 | 1
Infections and infestations - Other, unspecified (Infections and infestations) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panobinostat 20 mg (N=10) | Panobinostat 30 mg (N=16)
Platelet Count Decreased (Investigations) | 6 | 15
Anemia (Blood and lymphatic system disorders) | 7 | 12
Fatigue (General disorders) | 7 | 12
Neutrophil Count Decreased (Investigations) | 4 | 15
Diarrhea (Gastrointestinal disorders) | 8 | 8
Anorexia (Metabolism and nutrition disorders) | 2 | 12
Nausea (Gastrointestinal disorders) | 6 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 3
White Blood Cell Decreased (Investigations) | 2 | 8
Dizziness (Nervous system disorders) | 5 | 4
Edema (General disorders) | 3 | 5
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 3 | 5
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Fever (General disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 3 | 3
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 5
Constipation (Gastrointestinal disorders) | 1 | 3
Dysgeusia (Nervous system disorders) | 2 | 2
Gastrointestinal Disorders - Other, Stomatitis (Gastrointestinal disorders) | 1 | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Non-Cardiac Chest Pain (General disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Bruising (Injury, poisoning and procedural complications) | 0 | 3
Cardiac Disorders - Other, Systolic Murmur (Cardiac disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 1
Electrocardiogram Qt Corrected Interval Prolonged (Cardiac disorders) | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
General Disorders And Administration Site Conditions - Other, Pain At Port Site (General disorders) | 3 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1
Skin And Subcutaneous Tissue Disorders - Other, Ecchymosis (Skin and subcutaneous tissue disorders) | 3 | 0
Cardiac Disorders - Other, Tachycardia (Cardiac disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 0
Hematoma (Vascular disorders) | 2 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Respiratory, Thoracic And Mediastinal Disorders - Other, Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Skin And Subcutaneous Tissue Disorders - Other, Petechiae (Skin and subcutaneous tissue disorders) | 1 | 1
Skin Infection (Infections and infestations) | 1 | 1
Upper Respiratory Infection (Infections and infestations) | 1 | 1
Urinary Frequency (Renal and urinary disorders) | 1 | 1
Weight Loss (Investigations) | 0 | 1

LIMITATIONS AND CAVEATS:
Results of a planned interim analysis demonstrated that the regimen did not demonstrate sufficient evidence of efficacy necessary to justify further enrollment. Per protocol, the results of this analysis led to early termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.